CLINICAL TRIAL: NCT00335764
Title: Phase I/II Studies of BAY 43-9006 (Sorafenib) in Combination With OSI-774 (Erlotinib), R115777 (Tipifarnib) or CCI-779 (Temsirolimus) in Patients With Recurrent Glioblastoma Multiforme or Gliosarcoma
Brief Title: Sorafenib Combined With Erlotinib, Tipifarnib, or Temsirolimus in Treating Patients With Recurrent Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00676; NCI-2009-00676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000476286; NABTC-05-02 (Other: Adult Brain Tumor Consortium); NABTC-05-02 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Sorafenib; Erlotinib Hydrochloride; tipifarnib; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Patients receive oral sorafenib tosylate twice daily and oral erlotinib hydrochloride once daily on days 1-28.
  Interventions: Drug: sorafenib tosylate; Drug: erlotinib hydrochloride
- Group 2 (Experimental): Patients receive sorafenib tosylate as in group 1. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: sorafenib tosylate; Drug: temsirolimus
- Group 3 (Experimental): Patients receive sorafenib tosylate as in group 1. Patients also receive oral tipifarnib twice daily on days 1-21.
  Interventions: Drug: sorafenib tosylate; Drug: tipifarnib

INTERVENTIONS:
Drug: sorafenib tosylate — given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: erlotinib hydrochloride — given orally
  Other Names: CP-358,774; erlotinib; OSI-774
  Arms: Group 1
Drug: tipifarnib — given orally
  Other Names: R115777; Zarnestra
  Arms: Group 3
Drug: temsirolimus — IV administration
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
  Arms: Group 2

SUMMARY:
This phase I/II trial is studying the side effects and best dose of erlotinib, tipifarnib, and temsirolimus when given together with sorafenib and to see how well they work in treating patients with recurrent glioblastoma multiforme or gliosarcoma. Sorafenib, erlotinib, tipifarnib, and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib and tipifarnib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib together with erlotinib, tipifarnib, or temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase 1

1. Determine the maximum tolerated dose (MTD) of tipifarnib, erlotinib hydrochloride, or temsirolimus in combination with a fixed dose of sorafenib in patients with recurrent glioblastoma multiforme or gliosarcoma who are not taking enzyme-inducing antiepileptic drugs.

SECONDARY OBJECTIVES:

Phase 1 and 2

1. Characterize the safety profile of the doublet combinations of tipifarnib-sorafenib, erlotinib hydrochloride-sorafenib, and temsirolimus-sorafenib in patients with recurrent glioblastoma multiforme or gliosarcoma.
2. Characterize the pharmacokinetics of these doublet combinations, evaluating single-agent pharmacokinetics of each agent and the combination pharmacokinetics to determine drug-drug interactions.

Phase 2

1. Determine the efficacy of each of the doublet combinations, in terms of 6-month progression-free survival, in patients with recurrent glioblastoma multiforme or gliosarcoma.
2. Determine the efficacy of each of the doublet combinations, in terms of 12-month survival and objective tumor response, in patients with recurrent glioblastoma multiforme or gliosarcoma.

TERTIARY OBJECTIVES:

Phase 2

1. Perform exploratory correlative laboratory studies by examining tissue markers of signal transduction pathways by immunohistochemical analysis using tissue blocks obtained prior to initiation of protocol therapy, either from the time of diagnosis or subsequent tumor resection.
2. Determine the relationship between tumor and blood biomarkers and clinical outcome of patients treated with the combination of targeted agents.

OUTLINE:

This is a multicenter, phase I, dose-escalation study of tipifarnib, erlotinib hydrochloride, and temsirolimus followed by a phase II open-label study.

PHASE I:

Patients are sequentially assigned to 1 of 3 treatment groups.

GROUP 1: Patients receive oral sorafenib twice daily and oral erlotinib hydrochloride once daily on days 1-28.

GROUP 2: Patients receive sorafenib as in group 1. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.

GROUP 3: Patients receive sorafenib as in group 1. Patients also receive oral tipifarnib twice daily on days 1-21.

In all groups, treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

In each treatment group, cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride (group 1), temsirolimus (group 2), or tipifarnib (group 3) sequentially until the maximum tolerated dose (MTD) is determined for each group. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course of therapy.

PHASE II:

Patients receive sorafenib as in phase I. Patients also receive erlotinib hydrochloride, temsirolimus, or tipifarnib as in phase I at the MTD determined in phase I.

Tissue that was collected during a prior surgery is examined for biomarkers by immunohistochemistry (in patients enrolled in the phase II portion of the study). Biomarkers examined include epidermal growth factor receptor, Receptor tyrosine-protein kinase (HER-2), Protein kinase B (AKT), S6 ribosomal protein, and Receptor-linked tyrosine kinases (Erk).

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial glioblastoma multiforme or gliosarcoma
* Evidence of tumor progression by MRI or CT scan within the past 14 days AND on a steroid dose that has been stable for ≥ 5 days
* Patients who underwent prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis by either positron emission tomography or thallium scanning, magnetic resonance (MR) spectroscopy, or surgical documentation of disease
* Recent resection of recurrent or progressive tumor allowed
* Residual disease is not required
* Treatment for any number of prior relapses, defined as disease progression after initial therapy (i.e., radiotherapy with or without chemotherapy if used as initial treatment), allowed (phase I)
* No more than 3 prior therapies (initial therapy and therapy for 2 relapses) (phase II)
* Each of the following is considered 1 relapse:

  * Disease progression after initial therapy (i.e., radiotherapy with or without chemotherapy if used as initial therapy)
  * Underwent a surgical resection for relapsed disease and received no anticancer therapy for up to 12 weeks after surgical resection AND then underwent a subsequent surgical resection
  * Received prior therapy for a low-grade glioma, followed by a surgical diagnosis of glioblastoma
  * Failed prior radiotherapy
* 15 unstained paraffin slides or 1 tissue block must be available from original surgery, definitive surgery, or surgery closest to the initiation of this study (phase II)
* Karnofsky performance status 60-100%
* White Blood Cell (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin normal
* Creatinine < 1.5 mg/dL
* Prothrombin time (PT)/ international normalized ratio (INR) ≤ 1.5 (INR < 3.0 for patients on anticoagulation therapy)
* INR < 1.1 times upper limit of normal (ULN) (for patients on prophylactic anticoagulation therapy [low-dose warfarin])
* Fasting cholesterol < 350 mg/dL (for patients receiving temsirolimus and sorafenib)
* Fasting triglycerides < 400 mg/dL (for patients receiving temsirolimus and sorafenib)
* Well-controlled hypertension (e.g., systolic blood pressure ≤ 140 mm Hg or diastolic pressure ≤ 90 mm Hg) allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks (women) or 3 months (men) after completion of study treatment
* No peripheral neuropathy > grade 1 (for patients receiving sorafenib and tipifarnib)
* No evidence of bleeding diathesis or coagulopathy
* No history of any other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for ≥ 3 years
* No significant traumatic injury within the past 21 days
* No active infection or serious medical illness that would preclude study treatment
* No condition that would impair ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation or active peptic ulcer disease)
* No HIV disease
* No allergies to imidazoles (e.g., clotrimazole, ketoconazole, miconazole or econazole) or a history of allergic reactions attributed to any compound of similar chemical or biological composition to tipifarnib (for patients receiving sorafenib and tipifarnib)
* No other disease that would obscure toxicity or dangerously alter drug metabolism
* Recovered from prior therapy
* At least 7 days since prior noncytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin) (radiosensitizer does not count)
* At least 14 days since prior vincristine
* At least 21 days since prior procarbazine or major surgery
* At least 28 days since prior investigational agent or cytotoxic therapy
* At least 42 days since prior nitrosoureas or radiotherapy
* No prior sorafenib, AEE788, or vatalanib
* No prior surgical procedures affecting absorption
* No prior tipifarnib, lonafarnib, or other agents targeting farnesyl transferase (for patients receiving sorafenib and tipifarnib)
* No prior temsirolimus or mechanistic target of rapamycin (mTOR-targeting agent) (phase II), rapamycin or everolimus, or Akt-pathway inhibitors (for patients receiving sorafenib and temsirolimus)
* No prior erlotinib hydrochloride, multitargeted human epidermal receptor (AEE788), or other epidermal growth factor receptor targeting agents (phase II) (for patients receiving sorafenib and erlotinib hydrochloride)
* No concurrent enzyme-inducing antiepileptic drugs (e.g., carbamazepine, oxcarbazepine, phenytoin, fosphenytoin, phenobarbital, or primidone)
* Dexamethasone allowed
* No concurrent hepatic cytochrome p450 enzyme-inducing anticonvulsants
* No other concurrent investigational agents or anticancer therapies, including chemotherapy, radiotherapy, hormonal therapy, or immunotherapy
* No concurrent prophylactic filgrastim (G-CSF) or other hematopoietic colony-stimulating factors
* Full-dose anticoagulants allowed provided both of the following criteria are met:

  * In-range INR (between 2-3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-04; Primary Completion 2010-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gilbert, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - University of California at Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients enrolled from 2006 - 2009 Patients accrued from comprehensive outpatient cancer centers
Groups:
- Group 1 Phase I Sorafenib and Erlotinib: Patients receive oral sorafenib tosylate BID and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID (fixed) Dose Level 1: 400mg BID (fixed)
  erlotinib hydrochloride: given orally Dose Level 0: 100mg QD Dose Level 1: 100mg QD Dose Level 2: 150mg QD
- Group 2 Phase I Sorafenib and Temsirolimus: Patients receive sorafenib tosylate BID as in group 2. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID Dose Level 1: 400mg BID
  temsirolimus: IV administration Dose Level 0: 25mg IV QW Dose Level 1: 25mg IV QW Dose Level 2: 50mg IV QW Dose Level 3: 75mg IV QW Dose Level 4: 125mg IV QW Dose Level 5: 175mg IV QW
- Group 3 Phase I Sorafenib and Tipifarnib: Patients receive sorafenib tosylate BID as in group 3. Patients also receive oral tipifarnib twice daily on days 1-21.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID Dose Level 1: 400mg BID
  tipifarnib: given orally Dose Level 0: 100mg BID Dose Level 1: 100mg BID Dose Level 2: 200mg BID Dose Level 3: 300mg BID
- Group 1 Phase II Sorafenib and Erlotinib: Patients receive oral sorafenib tosylate BID and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally
  erlotinib hydrochloride: given orally
- Group 2 Phase II Sorafenib and Temsirolimus: Patients receive sorafenib tosylate BID as in group 2. Patients also receive temsirolimus IV 25 mg over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally 400mg BID
  temsirolimus: IV administration 25mg IV QW
Period: Overall Study
Arm/Group | Group 1 Phase I Sorafenib and Erlotinib | Group 2 Phase I Sorafenib and Temsirolimus | Group 3 Phase I Sorafenib and Tipifarnib | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Started | 17 | 13 | 24 | 19 | 19
Completed | 16 | 13 | 24 | 19 | 18
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — wrong histology | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: In Group 1 Phase 1 and Group 2 Phase 2 - each had a patient with wrong histology that made the patient ineligible and hence was not included in any of the analysis. Thus, total enrollment was 92 but only 90 evaluable patients
Groups:
- Group 1 Phase I Sorafenib and Erlotinib; Group 1 Phase II Sorafenib and Erlotinib: Patients receive oral sorafenib tosylate twice daily and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally
  erlotinib hydrochloride: given orally
- Group 2 Phase I Sorafenib and Temsirolimus: Patients receive sorafenib tosylate as in group 2. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally
  temsirolimus: IV administration
- Group 3 Phase I Sorafenib and Tipifarnib: Patients receive sorafenib tosylate as in group 3. Patients also receive oral tipifarnib twice daily on days 1-21.
  sorafenib tosylate: given orally
  tipifarnib: given orally
- Group 2 Phase II Sorafenib and Temsirolimus: Patients receive sorafenib tosylate 400 mg BID as in group 2. Patients also receive temsirolimus IV 25 mg over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally
  temsirolimus: IV administration
- Total: Total of all reporting groups
Arm/Group | Group 1 Phase I Sorafenib and Erlotinib | Group 2 Phase I Sorafenib and Temsirolimus | Group 3 Phase I Sorafenib and Tipifarnib | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus | Total
Number analyzed (Participants) | 16 | 13 | 24 | 19 | 18 | 90
Age, Continuous [Mean (Full Range); unit: years] | 53 [36 to 70] | 50 [32 to 59] | 57 [27 to 76] | 52 [30 to 76] | 50 [24 to 64] | 53 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 8 | 10 | 9 | 38
  Male | 9 | 9 | 16 | 9 | 9 | 52
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [70 to 100] | 80 [60 to 100] | 85 [60 to 100] | 90 [60 to 100] | 90 [60 to 100] | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of the Each Combination Agent Combined With a Fixed Dose of BAY 43-9006 Determined by Dose-limiting Toxicities (DLT) (Phase I)
Description: DLT defined as: any grade 4 hematologic toxicity; grade 3 thrombocytopenia > 7 days, any grade 3/4 non-hematologic toxicity (despite maximal medical therapy), any intolerable grade 2 non-hematological, ro grade 3 hematological toxicity requiring deduction during first 28 days of treatment, any toxicity resulting in delay of >1week during first 28 days of treatment
Time Frame: 28 days
Population: 3+3 design due to excessive toxicities of Group 3 no DLT was defined for Group 3
Measure: Number; unit: mg
Groups:
- Group 1 Phase I Sorafenib and Erlotinib QD: Patients receive oral sorafenib tosylate BID and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID (fixed) Dose Level 1: 400mg BID (fixed)
  erlotinib hydrochloride: given orally Dose Level 0: 100mg QD Dose Level 1: 100mg QD Dose Level 2: 150mg QD
- Group 2 Phase I Sorafenib and Temsirolimus QW: Patients receive sorafenib tosylate BID as in group 2. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID Dose Level 1: 400mg BID
  temsirolimus: IV administration Dose Level 0: 25mg IV QW Dose Level 1: 25mg IV QW Dose Level 2: 50mg IV QW Dose Level 3: 75mg IV QW Dose Level 4: 125mg IV QW Dose Level 5: 175mg IV QW
- Group 3 Phase I Sorafenib and Tipifarnib BID: Patients receive sorafenib tosylate BID as in group 3. Patients also receive oral tipifarnib twice daily on days 1-21.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID Dose Level 1: 400mg BID
  tipifarnib: given orally Dose Level 0: 100mg BID Dose Level 1: 100mg BID Dose Level 2: 200mg BID Dose Level 3: 300mg BID
Arm/Group | Group 1 Phase I Sorafenib and Erlotinib QD | Group 2 Phase I Sorafenib and Temsirolimus QW | Group 3 Phase I Sorafenib and Tipifarnib BID
Number analyzed (Participants) | 16 | 13 | 24
mg | 100 | 25 | NA — due to the excessive toxicities of Group 3 no DLT was defined

2. Primary Outcome: Pharmacokinetic Max Concentration (Cmax) of Group 2 Sorafenib and Temsirolimus (Phase I)
Description: Group 2: 13 patients received temsirolimus 25mg IV and 7 patients treated with 200mg Sorafenib and 6 patients treated with 400mg Sorafenib
Time Frame: cycle 1 ((Day1, Day15, Day28)
Population: Group 2: total 13 patients were studied for their day 1 Cmax ,day 15 Cmax and day 28 Cmax Note that although 13 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 2 Phase I Temsirolimus 25mg QW: Pt receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Patients receive sorafenib tosylate BID.
  sorafenib tosylate: given orally
  temsirolimus: IV administration 25mg
- Group 2 Phase I Sorafenib 200mg BID: Patients receive sorafenib tosylate BID 200mg. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally 200mg
  temsirolimus: IV administration 25mg
- Group 2 Phase I Sorafenib 400mg BID: Patients receive sorafenib tosylate BID 400mg. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally 400mg
  temsirolimus: IV administration 25mg
Arm/Group | Group 2 Phase I Temsirolimus 25mg QW | Group 2 Phase I Sorafenib 200mg BID | Group 2 Phase I Sorafenib 400mg BID
Number analyzed (Participants) | 13 | 7 | 6
ng/mL
  Day 1 Cmax | 530 (101) | NA (NA) — specimens not collected on day 1 | NA (NA) — specimens not collected on day 1
  Day 15 Cmax: number analyzed (Participants) | 12 | 4 | 4
  Day 15 Cmax | 616 (209) | 4.04 (1.68) | 7.49 (3.46)
  Day 28 Cmax: number analyzed (Participants) | 13 | 4 | 3
  Day 28 Cmax | NA (NA) — specimens not collected on day 28 | 3.26 (1.34) | 6.24 (4.03)

3. Primary Outcome: Pharmacokinetic cMax Group 1 Sorafenib and Erlotinib (Phase I)
Description: 8 samples collected over 24 hours on Day 1, day 15 and day 28
  13 total patients treated 100mg Erlotinib and either 200mg or 400mg of Sorafenib
Time Frame: 28days (D1, D15, D28) (0,1,2,4,6,8,12,24hr post administration)
Population: 8 samples collected over 24 hours on Day 1, day 15 and day 28 (0,1,2,4,6,8,12hr, & 24hr post administration). Note that although 16 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 1 Phase I Erlotinib 100mg QD: Patients receive oral oral erlotinib hydrochloride 100 mg once daily on days 1-28. Pts also receive Sorafenib tosylate BID
  sorafenib tosylate: given orally
  erlotinib hydrochloride: given orally
- Group 1 Phase I Sorafenib 200mg BID: Patients receive oral sorafenib tosylate BID 200mg oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally 200mg
  erlotinib hydrochloride: given orally
- Group 1 Phase I Sorafenib 400mg BID: Patients receive oral sorafenib tosylate BID 400mg and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally 400mg
  erlotinib hydrochloride: given orally
Arm/Group | Group 1 Phase I Erlotinib 100mg QD | Group 1 Phase I Sorafenib 200mg BID | Group 1 Phase I Sorafenib 400mg BID
Number analyzed (Participants) | 16 | 9 | 6
ng/mL
  cMax Day 1: number analyzed (Participants) | 14 | 9 | 6
  cMax Day 1 | 443 (155) | NA (NA) — Specimens not collected/drug not given on Day 1 | NA (NA) — Specimens not collected/drug not given on Day 1
  cMax Day 15 | 662 (373) | 5.51 (2.68) | 8.4 (5.18)
  cMax Day 28: number analyzed (Participants) | 10 | 7 | 3
  cMax Day 28 | 653 (469) | 4.67 (2.10) | 4.10 (0.56)

4. Primary Outcome: Pharmacokinetic AUC 0-12 Group 1 Sorafenib and Erlotinib (Phase I)
Description: 8 samples collected over 24 hours on Day 1, day 15 and day 28
  16 patients Note that although 16 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference AUC - Area Under Curve
Time Frame: 28Days (D1, D15, D28) (0,1,2,4,6,8,12,24hr post administration) AUC 0-12
Population: 8 samples collected over 24 hours on Day 1, day 15 and day 28 AUC 0-12 16 patients treated at 100mg erlotinib,and Sorafenib at either 200 or 400mg Note that although 16 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
Measure: Mean (Standard Deviation); unit: ug xhr/mL
Groups:
- Group 1 Phase I Erlotinib 100mg QD: Patients receive oral erlotinib hydrochloride 100 mg once daily on days 1-28.And also oral sorafenib tosylate BID
  sorafenib tosylate: given orally
  erlotinib hydrochloride: given orally
- Group 1 Phase I Sorafenib 200mg: Patients receive oral sorafenib tosylate BID 200mg and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally 200mg
  erlotinib hydrochloride: given orally
- Group 1 Phase I Sorafenib 400mg: Patients receive oral sorafenib tosylate BID 400mg and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally 400mg
  erlotinib hydrochloride: given orally
Arm/Group | Group 1 Phase I Erlotinib 100mg QD | Group 1 Phase I Sorafenib 200mg | Group 1 Phase I Sorafenib 400mg
Number analyzed (Participants) | 16 | 9 | 6
ug xhr/mL
  AUC0-12 Day1: number analyzed (Participants) | 14 | 9 | 6
  AUC0-12 Day1 | 6.3 (2.61) | NA (NA) — Specimens not collected/drug not given on Day 1 | NA (NA) — Specimens not collected/drug not given on Day 1
  AUC0-12 Day 15: number analyzed (Participants) | 6 | 9 | 5
  AUC0-12 Day 15 | 6.9 (4.59) | 45.85 (21.5) | 62.4 (38)
  AUC0-12 Day 28: number analyzed (Participants) | 8 | 7 | 3
  AUC0-12 Day 28 | 7.7 (4.05) | 40.29 (18.6) | 38.7 (9.61)

5. Primary Outcome: Trough Concentration Group 2 Sorafenib and Temsirolimus (Phase I)
Description: Group 2: 12 patients were analyzed for Day 1 (1 patient not evaluable), 5 patients were analyzed for Day 15 (8 patients not evaluable)
Time Frame: 15 days
Population: Group 2: 12 patients were analyzed for Day 1, 5 patients were analyzed for Day 15. In both cases samples were either missing or not enough to analyze.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 2 Phase I Sorafenib and Temsirolimus QW: Patients receive sorafenib tosylate BID Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally
  temsirolimus: IV administration
Arm/Group | Group 2 Phase I Sorafenib and Temsirolimus QW
Number analyzed (Participants) | 13
ng/mL
  Trough Day 1: number analyzed (Participants) | 12
  Trough Day 1 | 24 (6.92)
  Trough Day 15: number analyzed (Participants) | 5
  Trough Day 15 | 20 (7.05)

6. Primary Outcome: Plasma Time Curve (AUC) of Group 2 Sorafenib and Temsirolimus (Phase I)
Description: Day 1 = 12 patients (1 sample not evaluable) Day 15 = 5 patients (8 samples not evaluable)
  AUC - Area Under Curve
  8 samples collected over 24 hours - 28 day PKs
Time Frame: Cycle 1 (D1, D15, D28) (0,1,2,4,6,8,12,24hr post drug administration)
Population: 13 patients temsirolimus 25mg and Sorafenib at either 200mg or 400mg. 1 patient withdrew early hence specimens not analyzed in other cases samples were either missing or not enough to analyze if numbers are not 12
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Groups:
- Group 2 Phase I Temsirolimus 25mg QW: Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive sorafenib tosylate BID
  sorafenib tosylate: given orally Dose Level 0: 200mg BID Dose Level 1: 400mg BID
  temsirolimus: IV administration Dose Level 0: 25mg IV QW Dose Level 1: 25mg IV QW
- Group 2 Phase I Sorafenib 200mg: Patients receive sorafenib tosylate BID Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  temsirolimus: IV administration Dose Level 0: 25mg IV QW Dose Level 1: 25mg IV QW
- Group 2 Phase I Sorafenib 400mg: Patients receive sorafenib tosylate BID Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally Dose Level 1: 400mg BID
  temsirolimus: IV administration Dose Level 0: 25mg IV QW Dose Level 1: 25mg IV QW
Arm/Group | Group 2 Phase I Temsirolimus 25mg QW | Group 2 Phase I Sorafenib 200mg | Group 2 Phase I Sorafenib 400mg
Number analyzed (Participants) | 13 | 13 | 13
mcg*hr/mL
  AUC 0-12 Day 1: number analyzed (Participants) | 12 | 13 | 13
  AUC 0-12 Day 1 | 1.53 (0.27) | NA (NA) — Samples not collected on this day, drug not given on day 1 | NA (NA) — Samples not collected on this day, drug not given on day 1
  AUC 0-12 Day 15: number analyzed (Participants) | 5 | 3 | 1
  AUC 0-12 Day 15 | 1.35 (0.28) | 35.45 (18.10) | 42.32
  AUC 0-12 Day 28: number analyzed (Participants) | 13 | 13 | 2
  AUC 0-12 Day 28 | NA (NA) — Samples not collected on this day, drug not given on day 28 | 29.0 (12.32) | 32.98 (0.318)

7. Primary Outcome: Pharmacokinetic Cpmax Group 3 Sorafenib and Tipifarnib (Phase I) 100 mg QD (Level -1)
Description: Group 3: Only PKs for Dose level 1 and -1 were collected.
Time Frame: Cycle 1 = 28 day PKs D1, D15,D28 (0,1,2,4,6,8,12,24hr post drug administration)
Population: Group 3: Only PKs for Dose level 1 and -1 were collected. Note that although 6 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 3 Phase I Tipifarnib 100mg QD: Patients receive oral tipifarnib every day on days 1-21. Patients also receive sorafenib tosylate BID
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose level -1: 100mg QD
- Group 3 Phase I Sorafenib 200mg BID: Patients receive sorafenib tosylate BID Patients also receive oral tipifarnib every day on days 1-21.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose level -1: 100mg QD
Arm/Group | Group 3 Phase I Tipifarnib 100mg QD | Group 3 Phase I Sorafenib 200mg BID
Number analyzed (Participants) | 6 | 6
ng/mL
  Cmax Day 1: number analyzed (Participants) | 6 | 3
  Cmax Day 1 | 209.5 (135.85) | NA (NA) — Samples not collected on day 1, drug not given on day 1
  Cmax Day 15: number analyzed (Participants) | 6 | 3
  Cmax Day 15 | 169.5 (186) | 3.34 (1.31)
  Cmax Day 28 | NA (NA) — Samples not collected on day 28, drug not given on day 28 | 3.43 (1.46)

8. Primary Outcome: Pharmacokinetic CpMax Concentration of Group 3 Sorafenib and Tipifarnib (Phase I) 100mg BID
Description: Group 3: patients were studied for their day 1 Cmax, and day 15 Cmax Tipifanib and Day 15 and Day 28 sorafenib
  Group 3: Only PKs for Dose level 1 and -1 were collected.
Time Frame: Cycle 1 = 28 day PKs D1, D15,D28 (0,1,2,4,6,8,12,24hr post drug administration)
Population: Group 3: patients were studied for their day 1 Cmax, day 15 Cmax. and Day 28 Cmax PKs for 100mg BID Tipifarnib Note that although 10 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
  Level 1 (n=10): Day 1 n=6 (4 samples not evaluable) and D15 n=5 (5 samples not evaluable)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 3 Phase I Tipifarnib 100mg BID; Group 3 Phase I Sorafenib 200mg BID: Patients receive oral tipifarnib 100mg twice daily on days 2-21. Patients also sorafenib tosylate BID 200mg
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose Level 1: 100mg BID
Arm/Group | Group 3 Phase I Tipifarnib 100mg BID | Group 3 Phase I Sorafenib 200mg BID
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 1 Cmax: number analyzed (Participants) | 6 | 10
  Day 1 Cmax | 132.17 (65.96) | NA (NA) — Samples not collected on this day, drug not given
  Day 15 Cmax: number analyzed (Participants) | 5 | 5
  Day 15 Cmax | 233.60 (84.83) | 4.17 (2.99)
  Day 28 Cmax: number analyzed (Participants) | 10 | 7
  Day 28 Cmax | NA (NA) — Samples not collected on this day, drug not given | 4.53 (2.38)

9. Primary Outcome: Plasma Time Curve (AUC) of Group 3 Phase I Sorafenib and Tipifarnib 100mg QD (Level -1)
Description: Group 3: PKs for Dose level -1 100mg QD
  Note that although 9 patients were accrued/analyzed some samples were incomplete or inevaluable or missing hence number analyzed difference
Time Frame: Cycle 1 (D1, D15, D28) (0,1,2,4,6,8,12,24hr post drug administration)
Population: Group 3: PKs for Dose level -1 Tipifarnib 100mg QD Sorafenib started day 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Group 3 Phase I Tipifarnib 100mg QD: Patients receive oral tipifarnib 100mg twice daily on days 1-21. also receive sorafenib tosylate BID100mg
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose Level -1: 100mg QD
- Group 3 Phase I Sorafenib 200mg BID: Patients receive sorafenib tosylate BID100mgal and also tipifarnib 100mg QD on days 1-21.sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose Level -1: 100mg QD
Arm/Group | Group 3 Phase I Tipifarnib 100mg QD | Group 3 Phase I Sorafenib 200mg BID
Number analyzed (Participants) | 9 | 9
ng*hr/mL
  AUC 0-12 Day 1: number analyzed (Participants) | 6 | 9
  AUC 0-12 Day 1 | 814.5 (347.57) | NA (NA) — Samples not collected on this day, drug not given
  AUC 0-12 Day 15: number analyzed (Participants) | 2 | 3
  AUC 0-12 Day 15 | 706 (644.88) | 30.59 (14.59)
  AUC 0-12 Day 28 | NA (NA) — Samples not collected on this day, drug not given | 41.43 (28.82)

10. Primary Outcome: Plasma Time Curve (AUC) of Group 3 Phase I Sorafenib and Tipifarnib 100mg BID (Level 1)
Description: Group 3: PKs for Dose level 1 Tipifarnib 100mg BID
Time Frame: Cycle 1 = 28 day PKs D1, D15,D28 (0,1,2,4,6,8,12,24hr post drug administration)
Population: Group 3: PKs for Dose level 1 Tipifarnib 100mg BID
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Group 3 Phase I Tipifarnib 100mg QD: Patients receive oral tipifarnib twice daily on days 1-21. Patients also receive sorafenib tosylate BID 200 mg starting on day 2
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose Level 1: 100mg BID
- Group 3 Phase I Sorefenib 200mg BID: Patients also receive sorafenib tosylate BID 200 mg starting on day 2. Patients receive oral tipifarnib twice daily on days 1-21.
  sorafenib tosylate: given orally Dose Level 0: 200mg BID
  tipifarnib: given orally Dose Level 1: 100mg BID
Arm/Group | Group 3 Phase I Tipifarnib 100mg QD | Group 3 Phase I Sorefenib 200mg BID
Number analyzed (Participants) | 10 | 10
ng*hr/mL
  AUC 0-12 Day 1: number analyzed (Participants) | 6 | 10
  AUC 0-12 Day 1 | 631.67 (431.12) | NA (NA) — Samples not collected, drug not given on this day
  AUC 0-12 Day 15: number analyzed (Participants) | 4 | 2
  AUC 0-12 Day 15 | 390.25 (758.07) | 12.17 (16.33)
  AUC 0-12 Day 28: number analyzed (Participants) | 10 | 7
  AUC 0-12 Day 28 | NA (NA) — Samples not collected, drug not given on this day | 36.45 (17.21)

11. Primary Outcome: 12 Month Survival Rate (Phase II)
Description: number of patients alive at 12 months
Time Frame: 12 months
Population: Group 3 did not reach an MTD Hence, did not complete the Phase 2 portion of study, combination treatment too toxic.
Measure: Count of Participants; unit: Participants
Groups:
- Group 2 Phase II Sorafenib and Temsirolimus: Patients receive sorafenib tosylate BID as in group 2. Patients also receive temsirolimus IV 25 mg over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally
  temsirolimus: IV administration
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Number analyzed (Participants) | 19 | 18
Participants
  Patients Alive at 12 Months | 8 | 10
  Patients Dead at 12 Months | 11 | 8

12. Primary Outcome: Number of High Grade (3 and 4) Related Adverse Events of Each Combination Agent Combined With BAY 43-9006 (Phase I)
Description: CTCAE 3.0
Time Frame: 28 days
Measure: Number; unit: Events
Groups:
- Group 1 Phase I Sorafenib and Erlotinib QD: Patients receive oral sorafenib tosylate BID and oral erlotinib hydrochloride once daily on days 1-28.
  sorafenib tosylate: given orally
  erlotinib hydrochloride: given orally
- Group 2 Phase I Sorafenib and Temsirolimus QW: Patients receive sorafenib tosylate BID as in group 2. Patients also receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  sorafenib tosylate: given orally
  temsirolimus: IV administration
- Group 3 Phase I Sorafenib and Tipifarnib BID: Patients receive sorafenib tosylate BID as in group 3. Patients also receive oral tipifarnib twice daily on days 1-21.
  sorafenib tosylate: given orally
  tipifarnib: given orally
Arm/Group | Group 1 Phase I Sorafenib and Erlotinib QD | Group 2 Phase I Sorafenib and Temsirolimus QW | Group 3 Phase I Sorafenib and Tipifarnib BID
Number analyzed (Participants) | 16 | 13 | 24
Events
  Leukopenia Grade 3 | 0 | 0 | 0
  Lymphopenia Grade 3 | 0 | 2 | 3
  Neutropenia Grade 3 | 0 | 0 | 0
  Thrombocytopenia Grade 3 | 0 | 1 | 0
  AST, SGOT Grade 3 | 1 | 1 | 0
  Cholesterol Grade 3 | 0 | 1 | 0
  Diarrhea Grade 3 | 0 | 1 | 2
  Hemmorrhoids Grade 3 | 0 | 1 | 0
  Hypertriglyceridemia Grade 3 | 0 | 1 | 0
  Hypophosphatemia Grade 3 | 3 | 2 | 4
  Fatigue Grade 3 | 0 | 0 | 1
  Vomiting Grade 3 | 0 | 0 | 1
  Lipase Grade 4 | 0 | 0 | 3
  Joint - Knee Pain Grade 3 | 0 | 0 | 1
  Thrombosis/thrombus/embolism Grade 4 | 0 | 0 | 1
  Fever Grade 3 | 0 | 0 | 1
  Dysphasia Grade 3 | 0 | 0 | 1
  Pain - Head/Headache Grade 3 | 0 | 0 | 1
  Encephalopathy Grade 3 | 0 | 0 | 1
  Lipase Grade 3 | 1 | 0 | 0
  ALT, SGPT Grade 3 | 2 | 0 | 0
  Hypertension Grade 3 | 1 | 0 | 0

13. Primary Outcome: Number of High Grade (3 and 4) Related Adverse Events of Each Combination Agent Combined With BAY 43-9006 (Phase 2)
Time Frame: 1 year
Measure: Number; unit: events
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Number analyzed (Participants) | 19 | 18
events
  Lymphopenia Grade 3 | 2 | 2
  Thrombocytopenia Grade 3 | 0 | 5
  Thrombocytopenia Grade 4 | 0 | 2
  Cholesterol (high) Grade 3 | 0 | 2
  Diarrhea Grade 3 | 1 | 1
  Fatigue Grade 3 | 3 | 2
  Hypokalemia Grade 3 | 0 | 1
  Hyponatremia Grade 3 | 0 | 1
  Hypophosphatemia Grade 3 | 0 | 3
  Lipase (high) Grade 3 | 0 | 1
  Pharyngeal mucositis Grade 3 | 0 | 1
  Pruritis Grade 3 | 0 | 1
  Rash Grade 3 | 0 | 1
  Seizures Grade 3 | 0 | 1
  Hypertension Grade 3 | 1 | 0

14. Primary Outcome: Progression-free Survival at 6 Months (Phase II)
Description: Patients with a scan at 6 months without progressive disease Progressive disease defined as Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
Time Frame: 6 months
Population: Group 3 did not reach an MTD not complete the Phase 2 portion of study, combination treatment too toxic. End points not followed for group 3 Phase 2
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus | Group 3 Phase I Sorafenib and Tipifarnib BID
Number analyzed (Participants) | 19 | 18 | 24
weeks | 15.8 [3.4 to 39.6] | 8 [5 to 9] | 4.2 [0.1 to 21.1]

15. Primary Outcome: Objective Response Rate in Patients With Measurable Disease (Phase II)
Description: Measurable: Bidimensionally measurable lesions w/ clearly defined margins by MRI Evaluable: Unidimensionally measurable lesions, masses w/margins not clearly defined.
  Complete Response (CR): Complete disappearance of all measurable/evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients on minimal/no steroids.
  Partial Response (PR): >/= to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. Responders must be on same/decreasing doses of dexamethasone.
  Stable/No Response: Does not qualify for CR, PR, or progression. Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over BL if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Number analyzed (Participants) | 19 | 18
Participants
  Partial Response | 0 | 2
  Complete Response | 0 | 0
  Stable Response | 7 | 3
  Progressive Disease | 10 | 13
  Unevaluable | 2 | 0

16. Other Pre Specified Outcome: Exploratory Correlative Laboratory Studies (Phase II)
Description: Examination of tissue markers of signal transduction pathways by immunohistochemical analysis this was an exploratory measure and it was not explore due to the negative results of the rest of the study
Time Frame: 28 days
Population: this was more an exploratory correlative and as per the pre-specified protocol, was only to be performed if the outcome of other parts of the study indicated positive results.
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Molecular Targeted Combinations Correlative Study Initiative
Description: Determine the relationship between tumor and blood biomarkers and clinical outcome of patients this was more an exploratory correlative and was not completed due to the negative outcome of other parts of the study
Time Frame: 28 days
Population: as for outcome 16
Arm/Group | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: CTCAE
Arm/Group | Group 1 Phase I Sorafenib and Erlotinib | Group 2 Phase I Sorafenib and Temsirolimus | Group 3 Phase I Sorafenib and Tipifarnib | Group 1 Phase II Sorafenib and Erlotinib | Group 2 Phase II Sorafenib and Temsirolimus
All-Cause Mortality (participants affected / at risk) | 15/16 | 13/13 | 24/24 | 19/19 | 18/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13 | 4/24 | 1/19 | 2/18
Other Adverse Events (participants affected / at risk) | 13/16 | 8/13 | 15/24 | 11/19 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Phase I Sorafenib and Erlotinib (N=16) | Group 2 Phase I Sorafenib and Temsirolimus (N=13) | Group 3 Phase I Sorafenib and Tipifarnib (N=24) | Group 1 Phase II Sorafenib and Erlotinib (N=19) | Group 2 Phase II Sorafenib and Temsirolimus (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancrease infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Phase I Sorafenib and Erlotinib (N=16) | Group 2 Phase I Sorafenib and Temsirolimus (N=13) | Group 3 Phase I Sorafenib and Tipifarnib (N=24) | Group 1 Phase II Sorafenib and Erlotinib (N=19) | Group 2 Phase II Sorafenib and Temsirolimus (N=18)
Acidosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 7 (7) | 6 (6) | 3 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Lipase increased (Investigations) | 5 (5) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 5 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 3 (3)
Serum amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 6 (6) | 3 (3) | 3 (3) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to combo toxicities for Sorafenib and Tipifarnib exceeding monotherapy for each, MTD was not determined nor was Phase 2 explored.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less